CLINICAL TRIAL: NCT07255469
Title: Parameters Associated With Metabolic Response to Volume Expansion in Children Post-operative of Cardiac Surgery
Brief Title: Metabolic Fluid Responsiveness in Children
Acronym: METAFRIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/87; 2024-A02561-46 (Other: ID-RCB number)
Record Dates: First submitted 2025-09-01; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Circulatory Failure / Shock State; Fluid Therapy
Keywords: Circulatory failure; Critical Care; Echocardiography; Fluid therapy; Fluid responsiveness; Goal-directed fluid management; oxygen consumption; pediatrics; volume expansion
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to validate markers of metabolic fluid-responsiveness in children with acute circulatory failure following cardiac surgery. This would allow physicians to identify which patient could benefit the most from fluid expansion, thus avoiding useless and potentially dangerous fluid expansions that could lead to fluid overload. To this end, The investigators will evaluate the diagnostic accuracy of the ratio of central venous to arterial carbon dioxide tension (Pv-aCO2) to arteriovenous oxygen content (CavO2), a simple biological marker of anaerobic metabolism, for the diagnosis of metabolic fluid responsiveness defined as a significant increase in oxygen consumption (VO2) after fluid expansion.

DETAILED DESCRIPTION:
Acute circulatory failure, defined as a mismatch between oxygen delivery and consumption, is a frequent but serious condition in children after cardiac surgery. Fluid expansion is the cornerstone of acute circulatory failure treatment, but several studies have highlighted the adverse effects of excessive fluid expansion. Therefore, it is crucial to assess the individual benefit-risk ratio before each fluid expansion. Currently, finding fluid responsiveness tests is a major issue in intensive care. Usually, fluid responsiveness is defined as a significant improvement in stroke volume after fluid expansion. However, this is an intermediate objective, as the ultimate goal of the treatment is to restore an adequate balance between oxygen delivery and consumption. In adults, a significant proportion of hemodynamically successful volume expansions (i.e. resulting in a significant increase in stroke volume) are in fact metabolically ineffective, as they do not result in a significant increase in VO2. Certain biological parameters indicating anaerobiosis, such as the Pv-aCO2/CavO2 ratio, could be predictive of metabolic fluid responsiveness (e.g. a significant increase in VO2) in these patients. This has never been investigated in children.

The main objective of this study will be to evaluate the diagnostic accuracy of the Pv-aCO2/DAVO2 ratio at baseline for the diagnosis of metabolic fluid responsiveness, in children hospitalized in intensive care after cardiac surgery, for whom a fluid expansion was prescribed by the physician in charge.

The investigators will conduct a non-interventional, multicentric diagnostic accuracy study in French pediatric intensive care units. VO2 will be measured at baseline (e.g. before fluid expansion) and within 1h after fluid expansion by the combination of echocardiographic assessment and both arterial and venous blood gas. Blood gas are routinely measured, in patients already implanted with arterial and central line, to help manage acute circulatory failure. Echocardiography assessment, which is noninvasive and nonradiative, is also a common practice in this situation. Additional simple demographic, hemodynamic and clinical data will be collected at baseline and within 1 hour after fluid expansion, if monitored. No supplemental blood test or invasive parameter will be collected. These data will be collected from standard monitoring and/or from the patient's medical record.

The primary outcome is the diagnostic accuracy (measured by the area under the receiver operating characteristics curve) of the index test (Pv-aCO2/DAVO2 ratio at baseline) for the diagnostic of metabolic fluid responsiveness, defined as a 15% increase in VO2 after fluid expansion compared to baseline (gold standard test).

* VO2 (ml/min/m2) will be measured as follow, at baseline and within 1h after fluid expansion: VO2=(10.CO.DAVO2)/(Body Surface Area)
* DAVO2: difference between arterial and venous oxygen content (measured by blood gas analysis)
* CO: cardiac output, measured by transthoracic echocardiography as the product of heart rate, left ventricular outflow tract surface (from a parasternal long axis view) and left ventricular outflow tract velocity-time integral (from an apical 5-chambers view).

The secondary outcomes are:

* Diagnostic accuracy (AUROC, %) of the following index tests for the diagnosis of metabolic fluid responsiveness: arterial lactate, central venous oxygen saturation, Pv-aCO2.
* Association between fluid expansions induced tissular oxygen saturation variation and metabolic fluid responsiveness.
* Association between metabolic fluid responsiveness and hemodynamic profile (4 categories, depending on the increase of mean arterial pressure and/or stroke volume after fluid expansion)
* Subgroup analysis of the primary outcome: age, type of fluid expansion, circulatory physiology
* Association between baseline clinical data and metabolic fluid responsiveness Study design: non-interventional study of diagnostic accuracy (non-interventional, prospective, multi center). After a prescription of 10 ml/kg volume expansion by the physician in charge, screening for inclusion and exclusion criteria will be performed by an investigator physician. If the patient is included, volume expansion will be delayed for a few minutes (<5 min) while VO2 and the index test are measured. Within one hour after volume expansion, VO2 will be measured once again to evaluate the metabolic response to fluid expansion (gold-standard test).

Inclusion criteria: Age between 0 days and 15 years old; Patient hospitalized in an intensive care unit after cardiac surgery; Prescription of a 10ml/kg fluid expansion by the physician in charge; Prescription of arterial and venous blood gas before and after the volume expansion to help manage acute circulatory failure; Patient implanted with a functioning arterial line; Patient implanted with a functioning central venous line in the superior vena cava territory Exclusion criteria: Patient less than 37 weeks' corrected gestational age; Hemodynamic instability making the delay necessary for any test dangerous; Supine position contraindicated or deleterious; Impairment of echocardiographic acoustic window or restless patient making ultrasonography impossible; Opposition to participate expressed by the patient or by a parent or legal guardian Number of subjects: One hundred and ten patients are needed. This was calculated with the Obuchowski method, with an alpha risk of 0.05, a statistical power of 80%, a ratio "responder/non-responder" of 3, a predicted area under the receiver operating characteristics curve of 0.85 (based on previous studies) with a confidence interval greater than 0.75 which is a classic threshold for clinical pertinence.

Statistical analysis: Comparisons between metabolic "responders" and "non-responders" (to fluid expansion) will be performed with Student's t-test or Mann-Whitney test for continuous variables; or with the Chi-2 test or Fisher's exact test for categorical variables.

Metabolic fluid responsiveness represents the gold standard test. Patients will be classified as metabolic fluid responders in case of at least 15% increase in VO2 after fluid expansion, compared to baseline.

Diagnostic accuracy of the index tests will be explored. As multiple cut-offs of theses index tests can be defined, the investigators will report a receiver operating characteristic (ROC) curve which graphically represents the combination of sensitivity and specificity for each possible test positivity cut-off. The area under the ROC curve informs in a single numerical value about the overall diagnostic accuracy of the index test. The Youden index will also be calculated. The ROC curves of all index tests will be compared using a DeLong test.

A p value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 15 years old
* Hospitalization in a pediatric intensive care unit after cardiac surgery
* Prescription by the attending physician of a fluid expansion of 10ml/kg
* Prescription of arterial and venous blood gas before and after the volume expansion to help manage acute circulatory failure
* Patient implanted with a functioning arterial line
* Patient implanted with a functioning central venous line in the superior vena cava territory

Exclusion Criteria:

* Patient less than 37 weeks' corrected gestational age
* Hemodynamic instability making the delay necessary for any test dangerous
* Supine position contraindicated or deleterious
* Impairment of echocardiographic acoustic window or restless patient making ultrasonography impossible
* Opposition to participate expressed by the patient or by a parent or legal guardian

Ages: 0 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient hospitalized in an intensive care unit after cardiac surgery with a prescription of a 10ml/kg fluid expansion by the physician in charge
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-03-21 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUROC, %) of baseline Pv-aCO2/DAVO2 ratio to diagnose metabolic fluid | at baseline
  The primary outcome measure of a diagnostic accuracy study is the discriminative ability of an index test (expressed as an area under the ROC curve) to diagnose a condition (defined by a positive gold-standard reference test). In this study:
  * The index test is the baseline Pv-aCO2/DAVO2 ratio, i.e. the ratio between the veno-arterial carbon dioxide partial pressure gradient (mmHg) and the difference between arterial and venous oxygen content (ml.dl-1). Oxygen content and carbon dioxide partial pressure are measured by arterial and central venous blood gas analysis.
  * The condition is "metabolic fluid responsiveness"
  * The gold-standard reference test to diagnose metabolic fluid responsiveness is a VO2 increase of at least 15% between baseline and after volume expansion (i.e. ((VO2 after volume expansion - VO2 at baseline) / VO2 at baseline) > 15%). VO2 (ml/min/m2) will be measured as follow: VO2=(10.CO.DAVO2)/(Body Surface Area), where CO (ml.min-1) is the cardiac output, measured b

SECONDARY OUTCOMES:
AUROC (%) of the following index test to diagnose metabolic fluid responsiveness (same definition as above ) | at baseline
  Baseline arterial lactate (mmol.L-1), from an arterial blood gas analysis
AUROC (%) of the following index test to diagnose metabolic fluid responsiveness (same definition as above ) | at baseline
  Baseline central venous oxygen saturation (%), from a central venous blood gas analysis
AUROC (%) of the following index test to diagnose metabolic fluid responsiveness (same definition as above ) | at baseline
  Baseline Pv-aCO2 (mmHg), from an arterial and central venous blood gas analysis
Subgroup analysis of the primary outcome | at baseline
  age, type of fluid expansion, circulatory physiology
Correlation between metabolic fluid responsiveness and the following | at baseline
  * Age (0 - 2 years / 2 - 5 years / 5 - 15 years)
  * Sex
  * Weight
  * Number of fluid expansion during the last 24 h
  * Baseline Heart rate
  * Baseline arterial pressure
  * Baseline urine output
  * Baseline capillary refill time
  * Baseline mottling
  * Baseline left atrial pressure, if monitored as usual care
  * Baseline PELODS2 score
  * Type of volume expansion (albumin or crystalloid)
  * % of increase in cerebral near-infrared regional spectrophotometry (NIRS, %) ( baseline / after volume expansion)
  * % of increase in systemic near-infrared regional spectrophotometry (NIRS, %) ( baseline / after volume expansion)
  * % of increase in mean perfusion pressure (i.e. difference between mean arterial pressure and central venous pressure) ( baseline / after volume expansion)
  * % of increase in central venous pressure ( baseline / after volume expansion)
  * Hemodynamic profile
Correlation between metabolic fluid responsiveness and the following | at baseline , 28 days
  * Length of mechanical ventilation (days), evaluated 28 days after inclusion
  * Intensive care unit length of stay (days), evaluated 28 days after inclusion.
  * Mortality at 28 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Julien GOTCHAC, MD, Study Director — CHU de Bordeaux - Hôpital Cardiologique Haut Lévêque
Locations (8):
- France (8):
  - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron, France
  - Hôpital Jeanne de Flandre - CHU de Lille, Lille, France
  - Hôpital de la Timone - Assistance Publique - Hôpitaux de Marseille, Marseille, France
  - Hôpital mère-enfant - CHU de Nantes, Nantes, France
  - Hôpital Necker-Enfants Malades - Assistance Publique - Hôpitaux de Paris, Paris, France
  - Hôpital Cardiologique Haut Lévêque - CHU de Bordeaux, Pessac, France
  - Hôpital des enfants - CHU de Toulouse, Toulouse, France
  - Hôpital Felix Guyon - CHU de la Réunion, Saint-Denis, La Réunion